CLINICAL TRIAL: NCT04730973
Title: CARotid plaqUe StabilizatiOn and Regression With Evolocumab: the CARUSO Study
Brief Title: CARotid plaqUe StabilizatiOn and Regression With Evolocumab.
Acronym: CARUSO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Principal Investigator, Tiziana Claudia Aranzulla, MD, MSc, Azienda Ospedaliera Ordine Mauriziano di Torino
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-005663-31
Record Dates: First submitted 2021-01-24; First posted 2021-01-29 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab (Active Comparator): Subcutaneous evolocumab 140 mg will be administered every 2 weeks on top of optimal lipid-lowering therapy
  Interventions: Drug: Evolocumab; Other: lipid-lowering therapy (LLT)
- Standard (Placebo Comparator): No further treatment besides optimal lipid-lowering therapy will be administered
  Interventions: Other: lipid-lowering therapy (LLT)

INTERVENTIONS:
Drug: Evolocumab — Evolocumab 140 mg s.c. every two weeks on top of optimal lipid lowering therapy
  Other Names: Repatha
  Arms: Evolocumab
Other: lipid-lowering therapy (LLT) — lipid-lowering therapy (LLT)

SUMMARY:
The CARUSO trial aims at investigating the efficacy of evolocumab in promoting carotid plaque morphological stabilization and regression as compared to traditional lipid lowering therapy (LLT). Primary end-point of the study is the superiority of evolocumab on top of ongoing LLT versus ongoing LLT in carotid plaque morphological stabilization and regression at 6 and 12 months, respectively. Secondary end-points are: LDL-Cholesterol (LDL-C) absolute and percentage changes in the two groups at 12 month follow-up, and adverse cerebrovascular and cardiac events at 12 and 24 months

DETAILED DESCRIPTION:
Optimal lipid-lowering therapy (LLT) is a mainstay for the therapeutic management of atherosclerotic vascular disease. Cardiac and cerebrovascular adverse events and progression of atherosclerosis are, indeed, reduced in proportion to the achieved LDL cholesterol (LDL-C) levels.In addition, regression of atherosclerotic plaques with optimal LLT has been observed. However, optimal LLT with statin and ezetimibe, might be limited by the onset of adverse effects (i.e. disabling myalgias, diarrhea) with are usually dose -dependent, and the maximum tolerated statin dose might be insufficient to reach the recommended LDL-C goals. The advent of proprotein convertase subtilisin kexin type 9 inhibitors (PCSK9i) has allowed the achievement of very low LDL-C levels, and the fulfillment of the recommended LDL-C targets. However, while the experience with PCSK9i in patients with coronary artery disease has been wide, and coronary plaque regression has been documented, little is known regarding carotid plaque regression following therapy with PCSK9i. Only a few case reports have been published, and no observational study has been carried out so far. Furthermore, morphological carotid plaque stabilization has a prognostic role, and the possibility of its early achievement with PCSK9i may be relevant, especially in the context of percutaneous or surgical carotid interventions.

ELIGIBILITY:
Inclusion Criteria:

asymptomatic patients with uni- or bilateral carotid artery stenosis ≥50% and LDL-C values ≥100 mg/dL despite ongoing lipid lowering therapy

Exclusion Criteria:

* age <18 or ≥81 years old
* known intolerance to evolocumab
* ongoing or previous treatment with PCSK9i
* prior stroke or transient ischemic attack
* total carotid occlusion
* major active infection or major hematologic, renal, hepatic, or endocrine dysfunction
* malignancy with life expectancy below 24 months
* failure to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Morphological carotid plaque stabilization | Six months
  Morphological stabilization of the carotid plaque evaluated with Carotid duplex ultra-sonography
Carotid plaque regression | 12 months
  Carotid plaque regression evaluated with Carotid duplex ultra-sonography and defined as reduction of the entity of the stenosis and/or peak systolic velocity by at least 5%, as compared to baseline.

SECONDARY OUTCOMES:
Changes of LDL-C | 12 months
  Absolute changes of LDL-C
Major adverse cerebrovascular events | 12 and 24 months
  All-cause mortality, cardiovascular mortality, stroke, myocardial infarction, any coronary or peripheral revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Claudia Aranzulla, MD, Principal Investigator — A.O. Ordine Mauriziano di Torino
Locations (1):
- Azienda Ospedaliera Ordine Mauriziano di Torino, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aranzulla TC, Piazza S, Ricotti A, Musumeci G, Gaggiano A. CARotid plaqUe StabilizatiOn and regression with evolocumab: Rationale and design of the CARUSO study. Catheter Cardiovasc Interv. 2021 Jul 1;98(1):E115-E121. doi: 10.1002/ccd.29743. Epub 2021 Apr 24. PMID 33893754
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307